CLINICAL TRIAL: NCT03947983
Title: A Pilot Sensor-controlled Digital Gaming Intervention With Real-time Behavior Tracking to Motivate Self-management Behaviors in Older Adults With Heart Failure
Brief Title: Sensor-controlled Digital Game for Heart Failure Self-management
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Texas at Austin (Other)
Collaborators: National Institute of Nursing Research (NINR) (NIH)
Responsible Party: Principal Investigator, Kavita Radhakrishnan, Assistant Professor, University of Texas at Austin
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Supportive Care
Other Study IDs: 201800216-001; R21NR018229 (NIH)
Record Dates: First submitted 2019-05-08; First posted 2019-05-13 (Actual); Results first posted 2021-06-28 (Actual); Last update posted 2021-06-28 (Actual); Status verified 2021-06

CONDITIONS: Heart Failure
Keywords: self-management; digital game; sensor
MeSH Terms: conditions — Heart Failure

STUDY DESIGN:
Intervention Model Description: Participants will be randomized into two arms of intervention group or control group. The control group will receive only the weight monitoring and physical activity sensors while the intervention group will receive a sensor-controlled digital game (SCDG) app and weight monitoring and physical activity sensors
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention Group (Experimental): The intervention group will receive a sensor-controlled digital game (SCDG) app and weight monitoring and physical activity sensors
  Interventions: Behavioral: Sensor-controlled digital game (SCDG)
- Control group (Active Comparator): The control group will receive only the weight monitoring and physical activity sensors
  Interventions: Behavioral: Sensor Only

INTERVENTIONS:
Behavioral: Sensor-controlled digital game (SCDG) — The SCDG will involve a narrative, the goal of which is to help an avatar in the game avoid rehospitalization by using game points, earned via the participant's real-time behaviors, in game tasks that help maintain the avatar's optimal HF health status. Real-time behaviors of weight-monitoring and physical activity will be tracked by an off-the-shelf sensors and app (Withings). The data from the Withings sensors will then be routed to our SCDG app.
  The digital game paired with sensors will enable objective tracking of real-time behaviors such as physical activity, and weight monitoring, and provide personalized, contextually relevant feedback (e.g., reduce fluid intake or call doctor for weight gain) to motivate engagement in and generate habit formation of heart failure related self-management behaviors.
  Arms: Intervention Group
Behavioral: Sensor Only — Real-time behaviors of weight-monitoring and physical activity will be tracked by an off-the-shelf sensors and app (Withings). This group will also be provided with standardized evidence-based HF educational material.However, the data from the Withings sensors will not be routed to the SCDG.
  Arms: Control group

SUMMARY:
This study evaluates a sensor-controlled digital game (SCDG) to motivate self-management behaviors of weight monitoring and physical activity in older adults with heart failure (HF). Half of the participants will receive the SCDG app and weight monitoring and physical activity sensors and the other half will receive only the weight monitoring and physical activity sensors.

DETAILED DESCRIPTION:
The primary goal of this study is to obtain initial efficacy data and undertake a comprehensive feasibility assessment of a SCDG intervention that synchronizes with a Bluetooth-enabled weight scale and activity tracker to activate game rewards and feedback based on older adult heart failure (HF) participants' real-time weight monitoring and exercise behaviors.

The SCDG will involve a narrative, the goal of which is to help an avatar in the game avoid rehospitalization by using game points, earned via the participant's real-time behaviors, in game tasks that help maintain the avatar's optimal HF health status. Real-time behaviors of weight-monitoring and physical activity will be tracked by an off-the-shelf sensors and app (Withings). The data from the Withings sensors will then be routed to our SCDG app. The digital game paired with sensors will enable objective tracking of real-time behaviors such as physical activity, and weight monitoring, and provide personalized, contextually relevant feedback (e.g., reduce fluid intake or call doctor for weight gain) to motivate engagement in and generate habit formation of heart failure related self-management behaviors. The goal of this proposal is to demonstrate the feasibility of the SCDG concept with an optimal number of sensors in a small study so as to lay a foundation for scaling this concept to include more relevant sensors in longer, larger studies.

In this study, the initial efficacy of the SCDG intervention for primary outcome of rate of engagement in HF self-management behavior of weight-monitoring and secondary outcomes of physical activity engagement, HF self-management-knowledge, and self-efficacy, HF-functional status, hospitalization, cognitive ability, depression and quality of life will be evaluated. For this study, 44 older adults diagnosed with the New York Heart Association's HF classification I to III from out-patient HF settings in central Texas will be recruited, and randomized to either the SCDG intervention group that will receive sensors tracking weight monitoring and activity and play the SCDG on a mobile smartphone for 12 weeks or a control group that will receive sensors and an app tracking activity and weight monitoring, and standardized written HF educational modules.

ELIGIBILITY:
Inclusion Criteria:

* Age 55 years or older
* New York Heart Association (NYHA) heart failure classification of I to III that permits minimal physical activity without discomfort
* Understand English
* Pass a mini-cognitive screen
* Score of less than 2 (able to independently walk without using a cane or walker) on the Outcome and Assessment Information Set item for ambulation/locomotion
* Ownership of a smartphone or digital tablet

Exclusion Criteria:

* Severe visual (e.g., legally blind) or tactile (e.g., severe arthritis) impairments that adversely prevent the use of a smartphone or sensor devices
* History of renal failure which adversely affects heart failure prognosis
* Diagnosis of an end stage or terminal illness (e.g., cancer).

Min Age: 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 38 (Actual)
Dates: Start 2019-11-12 (Actual); Primary Completion 2020-11-10 (Actual); Study Completion 2021-01-30 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Kavita Radhakrishnan, PhD, Principal Investigator — The University of Texas Austin
Locations (2):
- United States (2):
  - Cardiac Floor, Seton Medical Center Austin, Austin, Texas
  - Cardiac Rehabilitation Center, Seton Medical Center Austin, Austin, Texas

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Radhakrishnan K, Julien C, Baranowski T, O'Hair M, Lee G, Sagna De Main A, Allen C, Viswanathan B, Thomaz E, Kim M. Feasibility of a Sensor-Controlled Digital Game for Heart Failure Self-management: Randomized Controlled Trial. JMIR Serious Games. 2021 Nov 8;9(4):e29044. doi: 10.2196/29044. PMID 34747701

RESULTS

PARTICIPANT FLOW:
Groups:
- Intervention Group: The intervention group will receive a sensor-controlled digital game (SCDG) app and weight monitoring and physical activity sensors
  Sensor-controlled digital game (SCDG): The SCDG will involve a narrative, the goal of which is to help an avatar in the game avoid rehospitalization by using game points, earned via the participant's real-time behaviors, in game tasks that help maintain the avatar's optimal heart failure (HF) health status. Real-time behaviors of weight-monitoring and physical activity will be tracked by an off-the-shelf sensors and app (Withings). The data from the Withings sensors will then be routed to our SCDG app.
  The digital game paired with sensors will enable objective tracking of real-time behaviors such as physical activity, and weight monitoring, and provide personalized, contextually relevant feedback (e.g., reduce fluid intake or call doctor for weight gain) to motivate engagement in and generate habit formation of heart failure related self-management behaviors.
- Control Group: The control group will receive only the weight monitoring and physical activity sensors
  Sensor Only: Real-time behaviors of weight-monitoring and physical activity will be tracked by an off-the-shelf sensors and app (Withings). This group will also be provided with standardized evidence-based heart failure (HF) educational material.However, the data from the Withings sensors will not be routed to the SCDG.
Period: Overall Study
Arm/Group | Intervention Group | Control Group
Started | 19 | 19
12 Weeks | 15 | 17
Completed (24 weeks) | 14 | 13
Not Completed | 5 | 6

BASELINE CHARACTERISTICS:
Groups:
- Intervention Group: The intervention group will receive a sensor-controlled digital game (SCDG) app and weight monitoring and physical activity sensors
  Sensor-controlled digital game (SCDG): The SCDG will involve a narrative, the goal of which is to help an avatar in the game avoid rehospitalization by using game points, earned via the participant's real-time behaviors, in game tasks that help maintain the avatar's optimal HF health status. Real-time behaviors of weight-monitoring and physical activity will be tracked by an off-the-shelf sensors and app (Withings). The data from the Withings sensors will then be routed to our SCDG app.
  The digital game paired with sensors will enable objective tracking of real-time behaviors such as physical activity, and weight monitoring, and provide personalized, contextually relevant feedback (e.g., reduce fluid intake or call doctor for weight gain) to motivate engagement in and generate habit formation of heart failure related self-management behaviors.
- Total: Total of all reporting groups
Arm/Group | Intervention Group | Control Group | Total
Number analyzed (Participants) | 19 | 19 | 38
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 11 | 9 | 20
  >=65 years | 8 | 10 | 18
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 10 | 10 | 20
  Male | 9 | 9 | 18
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 3 | 0 | 3
  Not Hispanic or Latino | 16 | 19 | 35
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 1 | 1
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 2 | 4 | 6
  White | 16 | 13 | 29
  More than one race | 1 | 1 | 2
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 19 | 19 | 38
Last heart failure hospitalization [Count of Participants; unit: Participants]
  < 6 months | 6 | 5 | 11
  7 months to 1 year | 2 | 3 | 5
  > 1 year | 11 | 11 | 22
Duration with heart failure diagnosis [Count of Participants; unit: Participants]
  < 30 days | 5 | 6 | 11
  1 month to 1 year | 8 | 5 | 13
  > 1 year | 6 | 8 | 14

OUTCOME MEASURES:

1. Primary Outcome: Number of Days With Weight-monitoring on Sensor Logs at 6 Weeks
Description: This outcome will be measured by collecting number of days with weight-monitoring data. This measure will be collected from sensor logs within the apps for both intervention group (IG) and control group (CG).
Time Frame: 6 weeks
Population: Based on participants available for data collection at 6 weeks.
Measure: Mean (Standard Deviation); unit: days
Arm/Group | Intervention Group | Control Group
Number analyzed (Participants) | 15 | 17
days | 35.8 (6.0) | 32.9 (10.5)

2. Primary Outcome: Number of Days With Weight-monitoring on Sensor Logs at 12 Weeks
Description: as for outcome 1
Time Frame: 12 weeks
Population: Based on participants available for data collection at 12 weeks.
Measure: Mean (Standard Deviation); unit: days
Arm/Group | Intervention Group | Control Group
Number analyzed (Participants) | 15 | 17
days | 69.7 (16.1) | 60.1 (18.7)

3. Secondary Outcome: Number of Days With Physical Activity on Sensor Logs at 6 Weeks
Description: This outcome measure will be measured by collecting number of days with physical activity data. These measures will be collected from sensor logs within the apps for both IG and CG.
Time Frame: 6 weeks
Population: Based on participants available for data collection at 6 weeks.
Measure: Mean (Standard Deviation); unit: Days
Arm/Group | Intervention Group | Control Group
Number analyzed (Participants) | 15 | 16
Days | 36.7 (10.9) | 39.2 (6.6)

4. Secondary Outcome: Number of Days With Physical Activity on Sensor Logs at 12 Weeks
Description: as for outcome 3
Time Frame: 12 weeks
Population: Based on participants available for data collection at 12 weeks.
Measure: Mean (Standard Deviation); unit: days
Arm/Group | Intervention Group | Control Group
Number analyzed (Participants) | 15 | 16
days | 76.6 (11.02) | 69.6 (17.3)

5. Secondary Outcome: Mean of Daily Steps on Physical Activity Sensor Logs at 6 Weeks
Description: This outcome measure will be measured by calculating the average daily steps at end of 6 weeks. These measures will be collected from sensor logs within the apps for both IG and CG.
Time Frame: 6 weeks
Population: Based on participants available for data collection at 6 weeks.
Measure: Mean (Standard Deviation); unit: steps
Arm/Group | Intervention Group | Control Group
Number analyzed (Participants) | 15 | 16
steps | 2742 (2499) | 2638 (1573)

6. Secondary Outcome: Mean of Daily Steps on Physical Activity Sensor Logs at 12 Weeks
Description: This outcome measure will be measured by calculating the average daily steps at end of 12 weeks. These measures will be collected from sensor logs within the apps for both IG and CG.
Time Frame: 12 weeks
Population: Based on participants available for data collection at 12 weeks.
Measure: Mean (Standard Deviation); unit: steps
Arm/Group | Intervention Group | Control Group
Number analyzed (Participants) | 15 | 16
steps | 2887 (2821) | 2541 (1604)

7. Secondary Outcome: Change From Baseline in Heart Failure Self-management Behaviors as Measured by the European Heart Failure Self-care Behavior Scale at 6 Weeks
Description: The instrument used will be 9-item European Heart Failure Self-care Behavior Scale (HSBS; standardized score from 0 to 100 (every item is given an equal weight) with a higher score meaning better self-care). Items are on a Likert scale of 1 - 5. For calculating the standardized score, each item is reverse coded and then computed using the formula: (Sum of all ever-coded items - 9)*2.7777
Time Frame: Baseline, 6 weeks
Population: Based on participants available for data collection for this measure at 6 weeks.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Intervention Group | Control Group
Number analyzed (Participants) | 15 | 15
score on a scale | 4.9 (20.4) | -2.7 (9.9)

8. Secondary Outcome: Change From Baseline in Heart Failure Self-management Behaviors as Measured by the European Heart Failure Self-care Behavior Scale at 12 Weeks
Description: The instrument used will be 9-item European Heart Failure Self-care Behavior Scale (HSBS; standardized score from 0 to 100 (every item is given an equal weight) with a higher score meaning better self-care. Items are on a Likert scale of 1 - 5. For calculating the standardized score, each item is reverse coded and then computed using the formula: (Sum of all ever-coded items - 9)*2.7777
Time Frame: Baseline, 12 weeks
Population: Based on participants available for data collection for this measure at 12 weeks.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Intervention Group | Control Group
Number analyzed (Participants) | 15 | 16
score on a scale | 9.3 (16.5) | 2.6 (12.4)

9. Secondary Outcome: Change From Baseline in Heart Failure Self-management Behaviors as Measured by the European Heart Failure Self-care Behavior Scale at 24 Weeks
Description: as for outcome 7
Time Frame: Baseline, 24 weeks
Population: Based on participants available for data collection for this measure at 24 weeks.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Intervention Group | Control Group
Number analyzed (Participants) | 12 | 13
score on a scale | 10.2 (13.4) | 0.5 (9.8)

10. Secondary Outcome: Change From Baseline in Heart Failure-related Quality of Life (QOL) on Kansas City Cardiomyopathy Questionnaire (KCCQ) at 6 Weeks
Description: The instrument used will be items 13 - 15 on the KCCQ. Values for the QoL domain range from 0 to 100 with higher scores indicating better quality of life. Domain score will be transformed to a 0 to 100 range by subtracting the lowest possible scale score, dividing by the range of the scale and multiplying by 100.
Time Frame: Baseline, 6 weeks
Population: Based on participants available for data collection for this measure at 6 weeks.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Intervention Group | Control Group
Number analyzed (Participants) | 14 | 16
score on a scale | 5.8 (13.1) | 8.7 (15.3)

11. Secondary Outcome: Change From Baseline in Heart Failure-related Quality of Life (QOL) on Kansas City Cardiomyopathy Questionnaire (KCCQ) at 12 Weeks
Description: as for outcome 10
Time Frame: Baseline, 12 weeks
Population: Based on participants available for data collection for this measure at 12 weeks.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Intervention Group | Control Group
Number analyzed (Participants) | 14 | 16
score on a scale | 8.2 (13.5) | 13.0 (19.3)

12. Secondary Outcome: Change From Baseline in Heart Failure-related Quality of Life (QOL) on Kansas City Cardiomyopathy Questionnaire (KCCQ) at 24 Weeks
Description: as for outcome 10
Time Frame: Baseline, 24 weeks
Population: Based on participants available for data collection for this measure at 24 weeks.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Intervention Group | Control Group
Number analyzed (Participants) | 13 | 13
score on a scale | 10.8 (16.9) | 15.4 (19.6)

13. Secondary Outcome: Change From Baseline in Heart Failure-related Functional Status on Kansas City Cardiomyopathy Questionnaire (KCCQ) at 6 Weeks
Description: The instrument used will be items 1-12 on the KCCQ. Values for the functional status summary score from 0 to 100 with higher scores indicating better quality of life. Summary score will be transformed to a 0 to 100 range by subtracting the lowest possible scale score, dividing by the range of the scale and multiplying by 100.
Time Frame: Baseline, 6 weeks
Population: Based on participants available for data collection for this measure at 6 weeks.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Intervention Group | Control Group
Number analyzed (Participants) | 14 | 16
score on a scale | 6.9 (14.1) | 1.7 (11.8)

14. Secondary Outcome: Change From Baseline in Heart Failure-related Functional Status on Kansas City Cardiomyopathy Questionnaire (KCCQ) at 12 Weeks
Description: as for outcome 13
Time Frame: Baseline, 12 weeks
Population: Based on participants available for data collection for this measure at 12 weeks.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Intervention Group | Control Group
Number analyzed (Participants) | 14 | 16
score on a scale | 3.7 (14.1) | 4.1 (12.6)

15. Secondary Outcome: Change From Baseline in Heart Failure-related Functional Status on Kansas City Cardiomyopathy Questionnaire (KCCQ) at 24 Weeks
Description: as for outcome 13
Time Frame: Baseline, 24 weeks
Population: Based on participants available for data collection for this measure at 24 weeks.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Intervention Group | Control Group
Number analyzed (Participants) | 13 | 13
score on a scale | 7.4 (10.7) | 6.5 (11.7)

16. Secondary Outcome: Number of Heart Failure Hospitalizations in the Past 6 Months at End of 24 Weeks as Assessed by Self-report
Description: This measure of number of cardiac hospitalizations in the past 6 months was obtained through participant self-report
Time Frame: Baseline, 24 weeks
Population: Based on participants available for data collection for this measure at 24 weeks.
Measure: Number; unit: hospitalizations
Arm/Group | Intervention Group | Control Group
Number analyzed (Participants) | 13 | 13
hospitalizations | 2 | 2

17. Secondary Outcome: Number of Heart Failure Hospitalizations in the Past Month at End of 12 Weeks as Assessed by Self-report
Description: This measure will be obtained through participant self-report
Time Frame: Baseline, 12 weeks
Population: Based on participants available for data collection for this measure at 12 weeks.
Measure: Number; unit: hospitalizations
Arm/Group | Intervention Group | Control Group
Number analyzed (Participants) | 15 | 16
hospitalizations | 0 | 1

18. Secondary Outcome: Number of Heart Failure Hospitalizations in the Past Month at End of 6 Weeks as Assessed by Self-report
Description: This measure will be obtained through participant self-report
Time Frame: Baseline, 6 weeks
Population: Based on participants available for data collection for this measure at 6 weeks.
Measure: Number; unit: hospitalizations
Arm/Group | Intervention Group | Control Group
Number analyzed (Participants) | 15 | 16
hospitalizations | 1 | 1

19. Secondary Outcome: Number of Heart Failure Hospitalizations in the Past Month at End of 24 Weeks as Assessed by Self-report
Description: This measure will be obtained through participant self-report
Time Frame: Baseline, 24 weeks
Population: Based on participants available for data collection for this measure at 24 weeks.
Measure: Number; unit: hospitalizations
Arm/Group | Intervention Group | Control Group
Number analyzed (Participants) | 13 | 13
hospitalizations | 1 | 0

20. Secondary Outcome: Change From Baseline in Heart Failure Self-management Knowledge on Atlanta Heart Failure Knowledge Test (AHKT) at 6 Weeks
Description: The instrument used will be 30-item Atlanta Heart Failure Knowledge Test (AHFKT). Each correct answer is scored as 1 point, with no additional weighting of items; correct responses are then summed. Incorrect or skipped questions are awarded 0 points. Total scores range from 0 to 30. Higher scores indicate better HF knowledge
Time Frame: Baseline, 6 weeks
Population: Based on participants available for data collection for this measure at 6 weeks.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Intervention Group | Control Group
Number analyzed (Participants) | 14 | 16
score on a scale | 1.9 (2.5) | 2.1 (2.5)

21. Secondary Outcome: Change From Baseline in Heart Failure Self-management Knowledge on Atlanta Heart Failure Knowledge Test (AHKT) at 12 Weeks
Description: as for outcome 20
Time Frame: Baseline, 12 weeks
Population: Based on participants available for data collection for this measure at 12 weeks.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Intervention Group | Control Group
Number analyzed (Participants) | 14 | 16
score on a scale | 1.4 (1.7) | 1.1 (1.5)

22. Secondary Outcome: Change From Baseline in Heart Failure Self-management Knowledge on Atlanta Heart Failure Knowledge Test (AHKT) at 24 Weeks
Description: as for outcome 20
Time Frame: Baseline,24 weeks
Population: Based on participants available for data collection for this measure at 24 weeks.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Intervention Group | Control Group
Number analyzed (Participants) | 12 | 13
score on a scale | 1.1 (2.1) | 1.1 (2.7)

23. Secondary Outcome: Change From Baseline in Heart Failure Self-efficacy on Self-efficacy Section of Self-care of Heart Failure Index at 24 Weeks
Description: The instrument used will be 6-item Section C Self-efficacy section of Self-care of heart failure Index (SCHFI). Scores on the self-efficacy scale will range from 0 to 100, with higher scores reflecting better self-efficacy. To standardize scores the formula: (sum of Section C items - 6) * 5.56 will be used.
Time Frame: Baseline, 24 weeks
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Intervention Group | Control Group
Number analyzed (Participants) | 12 | 13
score on a scale | 3.0 (18.0) | 7.0 (16.5)

24. Secondary Outcome: Change From Baseline in Heart Failure Self-efficacy on Self-efficacy Section of Self-care of Heart Failure Index at 12 Weeks
Description: as for outcome 23
Time Frame: Baseline, 12 weeks
Population: Based on participants available for data collection for this measure at 12 weeks.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Intervention Group | Control Group
Number analyzed (Participants) | 14 | 16
score on a scale | 1.0 (20.5) | 10.2 (12.3)

25. Secondary Outcome: Change From Baseline in Heart Failure Self-efficacy on Self-efficacy Section of Self-care of Heart Failure Index at 6 Weeks
Description: as for outcome 23
Time Frame: Baseline, 6 weeks
Population: Based on participants available for data collection for this measure at 6 weeks.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Intervention Group | Control Group
Number analyzed (Participants) | 14 | 16
score on a scale | 2.2 (25.7) | 6.9 (18.1)

26. Secondary Outcome: Change From Baseline in Relative Autonomy Index (RAI) as Measured on Treatment Self-Regulation Questionnaire (TSRQ) at 6 Weeks
Description: In the 19-item Treatment Self-Regulation Questionnaire (TSRQ) adapted for heart failure, each item can receive a value ranging from 1 - 7, as selected by the participant. The scale has 2 sub-scales: autonomous and controlled motivation. Calculating the scores for the sub-scales will consist of averaging the items on that subscale. They are:
  Autonomous Regulation: 2, 3, 7, 10, 13, 16, 18, 19. Scores for Autonomous Regulation can range from 8 to 56. High scores indicate high autonomous motivation or intrinsic motivation for behavior engagement.
  Controlled Regulation: 1, 4, 5, 6, 8, 9, 11, 12, 14, 15, 17. Scores for Controlled Regulation can range from 8 to 56. High scores indicate high controlled motivation or extrinsic motivation for behavior engagement.
  Scoring for RAI will consist of subtracting the average for Controlled Regulation from the average for Autonomous Regulation. Higher RAI scores indicate higher autonomous or intrinsic motivation for behavior engagement.
Time Frame: Baseline, 6 weeks
Population: Based on participants available for data collection for this measure at 6 weeks.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Intervention Group | Control Group
Number analyzed (Participants) | 14 | 17
score on a scale | -0.1 (1.2) | -0.2 (2.2)

27. Secondary Outcome: Change From Baseline in Relative Autonomy Index (RAI) as Measured on Treatment Self-Regulation Questionnaire (TSRQ) at 12 Weeks
Description: as for outcome 26
Time Frame: Baseline, 12 weeks
Population: Based on participants available for data collection for this measure at 12 weeks.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Intervention Group | Control Group
Number analyzed (Participants) | 14 | 17
score on a scale | 0.1 (2.6) | -0.3 (3.0)

28. Secondary Outcome: Change From Baseline in Relative Autonomy Index (RAI) as Measured on Treatment Self-Regulation Questionnaire (TSRQ) at 24 Weeks
Description: as for outcome 26
Time Frame: Baseline, 24 weeks
Population: Based on participants available for data collection for this measure at 24 weeks.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Intervention Group | Control Group
Number analyzed (Participants) | 13 | 13
score on a scale | -0.6 (2.5) | -0.2 (2.7)

ADVERSE EVENTS:
Time Frame: 24 weeks
Arm/Group | Intervention Group | Control Group
All-Cause Mortality (participants affected / at risk) | 0/19 | 0/19
Serious Adverse Events (participants affected / at risk) | 0/19 | 0/19
Other Adverse Events (participants affected / at risk) | 0/19 | 0/19

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol (2021-06-02): https://cdn.clinicaltrials.gov/large-docs/83/NCT03947983/Prot_000.pdf
  • Statistical Analysis Plan (2021-06-03): https://cdn.clinicaltrials.gov/large-docs/83/NCT03947983/SAP_001.pdf